CLINICAL TRIAL: NCT00067548
Title: A Phase 2 Study of EKB-569 in Subjects With Advanced Non-Small Cell Lung Cancer
Brief Title: Study Evaluating EKB-569 in Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3095A1-201
Record Dates: First submitted 2003-08-21; First posted 2003-08-25 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Non-Small-Cell Lung Carcinoma; Carcinoma, Non-Small Cell Lung; Lung Neoplasms
Keywords: Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — EKB 569

INTERVENTIONS:
Drug: EKB-569

SUMMARY:
This non-randomized, open-label, outpatient clinical trial is designed to assess the safety and efficacy of daily orally administered EKB-569 in subjects with advanced non-small cell lung cancer. Patients must have been previously treated with a platinum- and docetaxel-based therapy either given concurrently or as separate regimens.

The primary objective of the study is to assess the clinical activity of EKB-569 administered orally as a second-line or later stage treatment in subjects with advanced non-small cell lung cancer. Secondary objectives include:

* To further evaluate the safety of EKB-569
* To explore additional clinical activity parameters
* To explore subject survival
* To evaluate the pharmacokinetics of EKB-569
* To assess subject reported outcomes

EKB-569 will be administered orally as a single-agent. Eligible subjects will take EKB-569 daily as long as they do not have progressive disease and are tolerating treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated, institutional review board (IRB) or independent ethics committee (IEC)-approved informed consent form before any protocol-specific screening procedures
* Histologic and/or cytologic diagnosis of locally-advanced or metastatic non-small cell lung cancer in subjects who are not curable by conventional therapy

Exclusion Criteria:

* Chemotherapy, radiotherapy, anticancer immunotherapy, or investigational agents within 4 weeks of treatment day 1 (6 weeks if the previous regimen included mitomycin or nitrosoureas)
* Prior radiotherapy to >25% of bone marrow
* Prior epidermal growth factor receptor-targeting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer